CLINICAL TRIAL: NCT03826147
Title: Nitrite-boosting Therapy for Improving Physiological Function in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Douglas Seals, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 18-0364
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich beetroot juice (Active Comparator): Daily dose of nitrate-rich beetroot juice (70 mL) for 3 months.
  Interventions: Dietary Supplement: Nitrate-rich beetroot juice
- Nitrate-depleted beetroot juice (Placebo Comparator): Daily dose of nitrate-depleted beetroot juice (70 mL) for 3 months. The nitrate-depleted beetroot juice is identical in appearance, taste and caloric content to nitrate-rich beetroot juice, but with nitrate removed.
  Interventions: Dietary Supplement: Nitrate-depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Nitrate-rich beetroot juice — Daily supplementation with ~100 kcal of nitrate-rich beetroot juice containing 400 mg of dietary nitrate (James White Drinks, UK).
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Nitrate-depleted beetroot juice — Daily supplementation with ~100 kcal of nitrate-depleted beetroot juice (James White Drinks, UK).
  Arms: Nitrate-depleted beetroot juice

SUMMARY:
Nitric oxide (NO) is an essential molecule in the body that is decreased in patients with chronic kidney disease (CKD), leading to reductions in vascular, movement ("motor") and cognitive functions. This study will determine if daily oral supplementation (3 months) with a supplement that increases NO in the body, i.e., nitrate-rich beetroot juice, improves vascular, motor and cognitive function in patients with CKD; this study will also provide insight into the biological reasons (mechanisms) by which supplementation with nitrate-rich beetroot juice improves vascular function in these patients. Overall, this research will provide scientific evidence supporting the use of nitrate-rich beetroot juice for preserving physiological function and preventing co-morbid clinical conditions and disability in CKD.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage II-IV (eGFR using the Modification of Diet in Renal Disease (MDRD) prediction equation 20-90 mL/min/1.73m2; stable renal function in the past 3 months)
* Ability to give informed consent
* Albumin > 3.0 g/dL
* Ability to perform motor and cognitive tests (e.g., can rise from a chair, walk for 6 min, climb 10 stairs)
* Free from alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* Mini-mental state examination score >21 (rationale: to screen for subjects with major cognitive impairment)
* Blood pressure (BP) >100/60 mmHg for past 3 months (rationale: blood pressure below 100/60 mmHg may elevate the normally small risk of hypotension with nitrate supplementation)
* Not taking medications that will interfere with administered medications (e.g., sildenafil interacts with nitroglycerin)
* Body mass index (BMI) <40 kg/m2 (vascular function measurements can be inaccurate in severely obese patients)

Exclusion Criteria:

* Life expectancy <1 year
* Uncontrolled hypertension, defined as blood pressure > 160/100 mmHg in the past 3 months
* History of severe liver disease
* History of severe congestive heart failure (i.e., ejection fraction < 35%)
* History of hospitalizations within the last 3 months
* Active infection or antibiotic therapy
* Warfarin use
* Vasculitis requiring immunosuppressive therapy within the last year
* High dietary nitrate intake or current nitrate/nitrite supplementation; hypersensitivity to nitrates or nitrites
* Glucose-6-phosphate dehydrogenase deficiency or blood methemoglobin >2%
* Unwilling to abstain from use of mouthwash or other oral hygiene practices (e.g., tongue scraping) outside of teeth brushing that disrupt the oral microbiome and would interfere with nitrate conversion to nitrite
* Blood donation within 8 weeks prior to enrolling in the study; unwilling to abstain from donating blood for 8 weeks after completing the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in vascular endothelial function | Baseline, 3 months
  as measured by brachial artery flow-mediated dilation
Change in aortic stiffness | Baseline, 3 months
  as measured by carotid-femoral pulse wave velocity

SECONDARY OUTCOMES:
Change in oxidative stress-associated suppression of endothelial function assessed as the increase in brachial artery flow-mediated dilation following an ascorbic acid infusion | Baseline, 3 months
  The influence of oxidative stress on brachial artery flow-mediated dilation will be determined by infusing a supraphysiological dose of ascorbic acid known to scavenge superoxide or isovolumic saline
Change in endothelial cell markers of oxidative stress | Baseline, 3 months
  Endothelial cell nitrotyrosine levels will be determined

OTHER OUTCOMES:
Motor function composite score | Baseline, 3 months
  Multiple domains of motor function (including endurance, strength, dexterity) assessed using the NIH Toolbox Motor Battery (aggregated into one reported value)
Fluid cognition composite score | Baseline, 3 months
  Multiple domains of cognitive function (including executive function, memory, processing speed) assessed using the NIH Toolbox Cognitive Battery (aggregated into one reported value)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Rossman, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Integrative Physiology of Aging Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh ES, Opoku G, Darvish S, Craighead DH, Ostrow A, Rossman MJ, Steele CN, Struemph T, You Z, Seals DR, Chonchol M, Nowak KL. Sex Differences in Dementia and Mild Cognitive Impairment in Nondialysis CKD. Clin J Am Soc Nephrol. 2025 Nov 20. doi: 10.2215/CJN.0000000922. Online ahead of print. No abstract available. PMID 41264372
- [Derived] Jones AM, Vanhatalo A, Seals DR, Rossman MJ, Piknova B, Jonvik KL. Dietary Nitrate and Nitric Oxide Metabolism: Mouth, Circulation, Skeletal Muscle, and Exercise Performance. Med Sci Sports Exerc. 2021 Feb 1;53(2):280-294. doi: 10.1249/MSS.0000000000002470. PMID 32735111